

## Project Title:

A review of surgical management of Congenital Pulmonary Airway Malformations (CPAM): A decade of experience

## Institutions

Department of Anaesthesia Kings College Hospital, London.

Health Research Authority Approval

REC Reference: 18/NW/0294, IRAS Project ID: 238420

Correspondence

Chula Goonasekera <a href="mailto:chula.goonasekera@nhs.net">chula.goonasekera@nhs.net</a>

| (Parent name and address) |
|---|
| Dear |
| Requesting consent for a telephone interview (Hospital reference): |
| This is a letter of invitation for a research study. I am writing this letter expecting your participation as your child has undergone surgery to remove a lung lesion between 2007 and 2017 at xxx hospital. |
| We are currently reviewing all surgical and anaesthetic techniques used and the subsequent wellbeing of these children who underwent above surgery at Hospital xxx. The purpose is to understand their health, growth and development, post-surgery. This study is not an investigation of any medical concern. |
| Ms XYZ is a medical student gathering this information. She is hoping to submit her scientific findings and defend a thesis for her intercalated B Sc at ABC School of Medicine. |
| Should you give your consent, she shall telephone you at a convenient time of your choice indicated in the consent form (enclosed) returned completed. This 15-20-minute telephone interview is to understand your views on the benefits of surgery and your child's wellbeing, following his/her surgery. |
| Please reply using the stamped addressed envelope. Please also see attached patient information leaflet for more detail. |
| Your time and effort made on this contribution is most appreciated. |

Date: 24/04/2018

Yours truly,

## PARTICIPANT CONSENT FORM

| SHORT TITLE:<br>Surgical management of CPAM: a service and outcome review |
|---|
| FULL STUDY TITLE: A review of surgical management of Congenital Pulmonary Airway Malformations (CPAM): A decade of experience at a single centre, and patient outcomes |
| IRAS Number: 238420<br>Chief Investigator: Dr XXX : Consultant Anaesthetist |
| Participant Identification Number for this study: |
| Please initial box |
| 1 I confirm that I have read the information letter dated $02/11/2017$ (version.1.0) for the above study and the request for a telephone interview. |
| 2 I understand that my participation is voluntary and that I am free to withdraw at any time without giving any reason, without my legal rights being affected. |
| 3 I understand that relevant sections of my statements / recorded during the study, may be looked at by individuals from the sponsor of the trial (XXX Hospital) and responsible persons authorised by the sponsor, from regulatory authorities where it is relevant to my taking part in this research. I give permission for these individuals to have access to my / my child's records. |
| 4 I understand that the information collected about me/ my child will be used to support other research in the future, and may be shared anonymously with other researchers. |
| 5 I agree to take part in the above study and the telephone interview. |
| My most convenient time for a telephone interview shall be daytime 0900-1700/ evening 1700-2000/ or during the weekends 0900-1800/ (please delete as appropriate). |
| The telephone number/s that I am contactable are (please complete) |

(1) ......(2) ......(3) ......(3) .....

Name of Participant Date Signature